CLINICAL TRIAL: NCT03097237
Title: High Fiber Rye Foods for Weight and Body Fat Reduction
Acronym: RyeWeight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Responsible Party: Principal Investigator, Dr. Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SLU254
Record Dates: First submitted 2016-12-04; First posted 2017-03-31 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Wholegrain rye (Experimental): Wholegrain rye products with a high content of dietary fiber
  Interventions: Other: Wholegrain rye
- Refined wheat (Active Comparator): Refined wheat products with a low content of dietary fiber
  Interventions: Other: Refined wheat

INTERVENTIONS:
Other: Wholegrain rye — Cereal products based on wholegrain rye
  Arms: Wholegrain rye
Other: Refined wheat — Cereal products based on refined wheat
  Other Names: Control
  Arms: Refined wheat

SUMMARY:
The overall aim of this study is to investigate whether a diet rich in rye fiber from wholegrain rye, compared to refined wheat, as part of a hypocaloric diet leads to larger weight loss and lower body fat content after 12 weeks of intervention. Furthermore the study will investigate the effect on appetite as a potential underlying mechanism for differences in weight loss and body fat reduction.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-35 kg/m2
* Hb≥120g/l
* Serum thyroid stimulating hormone (TSH) ≤4.00 mIU/L
* Plasma low density lipoprotein cholesterol <5.3 mmol/L
* Plasma triglycerides ≤1.8 mmol/L
* Signed informed consent
* Freezer capacity for 2 weeks bread provision

Exclusion Criteria:

* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study
* Unable to complete satisfactorily the 3-day weighted food record at screening visit 2.
* Unable to lose 0.5 kg or more during the run-in period for men and women not having menstruation during the run in period
* Increased body weight, despite reported adherence to dietary intake for women with menstruation during the run-in period.
* Using nicotine products on a daily basis (incl. chewing gum, patches, snus etc.)
* Using e-cigarettes (regardless of nicotine content)
* Following any weight reduction program or having followed one during the last 6 months prior to visit 1
* Diastolic blood pressure 105 mm Hg at visit 1
* Systolic blood pressure 160 mm at visit 1
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* More than 10 hours physical activity per week
* History of heart failure or heart attack within 1 year prior to screening
* Have type I diabetes
* Receiving pharmacological treatment for type II diabetes (treatments based on life style interventions are acceptable, as long as they are compatible with the study protocol)
* Previous gastrointestinal surgery
* Thyroid disorder
* History of drug or alcohol abuse
* Stroke or transient ischemic attack (TIA) within 1 year prior to screening
* Consumption of drugs aimed at weight management or drugs affecting body weight to a degree that is considered unsuitable for study participation by responsible physician (will be included in the list of allowed/disallowed medications)
* Pregnant or lactating or wish to become pregnant during the period of the study.
* Food allergies or intolerances
* Vegetarian (due to the standardized meals for appetite measurements)
* Unable to understand written and spoken Swedish
* Lack of suitability for participation in the trial, for any reason, as judged by the medical doctor or PI.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Difference in body weight | 12 weeks
Difference in body fat mass | 12 weeks

SECONDARY OUTCOMES:
Appetite measured by visual analogue scale (VAS) questionnaire | 12 weeks
  Investigate if satiety differs between groups after 12 weeks of intervention and investigate if appetite correlates with changes in body weight. Measurements will be conducted through visual analogue scale (VAS) questionnaire, where participants log into a homepage and respond to their perceived satiety, hunger and desire to eat every 30-60 min during a day at base line, after 6w and 12wk.
Difference in body weight and body fat mass | 6 weeks
  Investigate if differences in body weight and body fat mass is evident already after 6 weeks
Fecal energy excretion by bomb calorimetry of 72h quantitative fecal collections. | 12 weeks
  Investigate differences in fecal energy excretion between the two intervention groups in a subgroup of 50 subjects. Every subject will be instructed to collect all feces in a special devise during 48h.
Gut microbiota | 6 and 12 weeks
Marker of glucose metabolism | 6 and 12 weeks
  Investigate differences in hemoglobin A1c (HbA1c)
Marker of Insulin resistance | 6 and 12 weeks
  Investigate differences in homeostatic model assessment insulin resistance (HOMA-IR)
Appetite regulation | 6 and 12 weeks
  Investigate differences in glucagon-like peptide 1(GLP-1)
Appetite | 6 and 12 weeks
  Investigate differences in leptin concentration
Marker of inflammation | 6 and 12 weeks
  Investigate differences in C-reactive protein (CRP).
Blood lipids | 6 and 12 weeks
  Investigate differences in triglyceride (TG), total cholesterol, high density lipoprotein(HDL) and low density lipoprotein (LDL).

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, Dr, Principal Investigator — Chalmers University of Technology
Locations (1):
- Chalmers University of Technology, Gothenburg, Sweden

REFERENCES:
- [Derived] Iversen KN, Carlsson F, Andersson A, Michaelsson K, Langton M, Riserus U, Hellstrom PM, Landberg R. A hypocaloric diet rich in high fiber rye foods causes greater reduction in body weight and body fat than a diet rich in refined wheat: A parallel randomized controlled trial in adults with overweight and obesity (the RyeWeight study). Clin Nutr ESPEN. 2021 Oct;45:155-169. doi: 10.1016/j.clnesp.2021.07.007. Epub 2021 Jul 24. PMID 34620312